CLINICAL TRIAL: NCT06412861
Title: Comparison of Propofol-ketamine and Propofol-fentanyl Sedation in Short-term Gynecological Cases
Brief Title: Propofol-ketamine or Propofol-fentanyl for Procedural Sedation in the Short-term Gynecological Case
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ilke
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Ketamine; Sedation; Gynecologic Disease
Keywords: ketamine; sedation; gynecological case
MeSH Terms: conditions — Genital Diseases, Female | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of two groups (1:1 ratio, parallel randomization) by randomization using the computer program "ResearchRandomizer" (Urbaniak and Plous 2013), conducted by a team member not involved in surgery or patient assessment. There will be 30 patients in each group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-propofol (Active Comparator): 0.5 mg/kg ketamine + 1 mg/kg propofol will be administered. Ramsey Sedation Score will be targeted to be > 4. For this, if necessary, additional iv 0.5 mg/kg propofol will be administered.
  Interventions: Drug: Ketamine
- fentanyl-propofol (Active Comparator): 1 mcg/kg fentanyl + 1 mg/kg propofol will be administered. Ramsay Sedation Score will be targeted to be > 4. For this, if necessary, additional iv 0.5 mg/kg propofol will be administered.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg ketamine + 1 mg/kg propofol, Ramsey Sedation Score > 4 will be targeted. For this, if necessary, additional iv 0.5 mg/kg propofol will be administered.
  Other Names: GROUP A
  Arms: ketamine-propofol
Drug: Fentanyl — 1 mcg/kg fentanyl + 1 mg/kg propofol will be administered. Ramsay Sedation Score will be targeted to be > 4. For this, if necessary, additional iv 0.5 mg/kg propofol will be administered.
  Other Names: GROUP B
  Arms: fentanyl-propofol

SUMMARY:
Comparison of fentanyl-propofol and ketamine-propofol combination for sedation in brief gynecological cases

Our study aimed to evaluate ketamine-propofol and fentanyl-propofol combinations in short-term gynecological cases in terms of hemodynamic parameters, recovery, complications, patient and physician comfort.

DETAILED DESCRIPTION:
Procedural sedation is widely used in various medical procedures worldwide, aiming to suppress consciousness adequately and provide sufficient analgesia while preserving the patient's cardiorespiratory function during painful or unpleasant interventions (1,2). Many drugs are used alone or in combination for this purpose (e.g., benzodiazepines, opioids such as fentanyl and remifentanil, midazolam, ketamine, propofol, dexmedetomidine) (6). This prospective, randomized, double-blind study will evaluate the effectiveness of ketamine-propofol and fentanyl-propofol combinations during short-term gynecological procedures by comparing the frequency of lower extremity movements in sedated patients.

Participants eligible for the study will include individuals aged 18-65 with American Society of Anesthesiologists (ASA) physical status I or II undergoing short gynecological procedures lasting less than 30 minutes. Participants with allergies to study medications, obesity, or behavioral disorders will be excluded. All participants will provide written informed consent the day before the procedure.

Enrolled participants will be divided into two groups: Group K, receiving ketamine and propofol, and Group F, receiving fentanyl and propofol. Heart rate (HR), arterial blood pressure (ABP), peripheral oxygen saturation (SpO2), Ramsey Sedation Score( 1: Awake; agitated or restless or both, 2: Awake; cooperative, oriented, and tranquil,3: Awake but responds to commands only, 4: Asleep; brisk response to light glabellar tap or loud auditory stimulus,5: Asleep; sluggish response to light glabellar tap or loud auditory stimulus, 6: Asleep; no response to glabellar tap or loud auditory stimulus)( RSS), and Facial Pain Score(0:No hurt- 10:Hurts worst (FPS) will be evaluated at five time points: T1 (pre-induction), T2 (1 minute post-induction), T3 (3 minutes post-induction), T4 (end of surgery), and T5 (30 minutes postoperatively).

) In Group K, ketamine-propofol will be prepared in a 1:1 ratio (both 10 mg/mL) in the same syringe, while in Group F, fentanyl (1-2 mcg/kg) and propofol (1 mg/kg) will be prepared separately. Sedation will be initiated with 0.2 mL/kg of ketofol. Surgery will commence if RSS > 4; if the desired sedation level is not achieved, a rescue dose of 0.5 mg/kg propofol bolus will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65,
* American Society of Anesthesiologists (ASA) I-II,

Exclusion Criteria:

* Patients with a known allergy to any of the drugs used in the study,
* Renal, hepatic, neuro-psychiatric, cardiovascular, or respiratory diseases, i
* intracranial space-occupying lesions,
* Pregnant women,
* Body mass index (BMI) > 30

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Surgical satisfaction | Postoperative procedure
  Surgical satisfaction survey:
  Was the level of sedation sufficient during local anesthesia administration? Was the level of sedation sufficient throughout the surgical procedure? Was your verbal communication level with the patient sufficient? Would you recommend this sedation method to other surgeons for this surgical procedure? Would you accept using the same sedation technique for your next surgical procedure with the patient? Scoring: Ratings are based on a scale of 0 to 2, where 0 indicates 'not at all', 1 indicates 'somewhat', and 2 indicates 'completely'. The scores are evaluated on a scale from the lowest '0' to the highest '10'."
Incidence of lower extremity movement during the procedure | intraoperative
  The incidence of lower extremity movement indicative of inadequate sedation or analgesia during the procedure

SECONDARY OUTCOMES:
Adverse events (such as nausea, vomiting, airway obstruction, apnea, desaturation, respiratory depression, hypotension and bradycardia) | 30th minute postoperative
  he side effects occurring during the intraoperative and postoperative periods include:
  Recall events (recall of events during surgery) Apnea (holding breath for >15 seconds) Desaturation (SpO2 < 96%) Jaw thrust maneuver Bradycardia (heart rate < 50 beats/min) Skin rash

CONTACTS AND LOCATIONS:
Overall Officials: ilke tamdoğan, Study Director — ndokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Sa Rego MM, Watcha MF, White PF. The changing role of monitored anesthesia care in the ambulatory setting. Anesth Analg. 1997 Nov;85(5):1020-36. doi: 10.1097/00000539-199711000-00012. No abstract available. PMID 9356094
- [Background] Badrinath S, Avramov MN, Shadrick M, Witt TR, Ivankovich AD. The use of a ketamine-propofol combination during monitored anesthesia care. Anesth Analg. 2000 Apr;90(4):858-62. doi: 10.1097/00000539-200004000-00016. PMID 10735789